CLINICAL TRIAL: NCT03127384
Title: A Randomised, Evaluator-blind Comparative Study to Evaluate Performance and Safety of Restylane Lidocaine and No-treatment Control for Treatment of Depressed Facial Acne Scars
Brief Title: Performance and Safety of Restylane Lidocaine for Treatment of Depressed Facial Acne Scars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 05DF1605
Record Dates: First submitted 2017-04-20; First posted 2017-04-25 (Actual); Results first posted 2019-10-03 (Actual); Last update posted 2022-08-26 (Actual); Status verified 2019-09

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No-treatment control (Experimental)
  Interventions: Other: No-treatment control
- Treatment (Experimental): Intradermal injection Restylane Lidocaine
  Interventions: Device: Restylane Lidocaine

INTERVENTIONS:
Device: Restylane Lidocaine — Hyaluronic acid based filler
  Arms: Treatment
Other: No-treatment control — No-treatment control
  Arms: No-treatment control

SUMMARY:
The purpose of this study is to evaluate performance and safety of Restylane Lidocaine for treatment of depressed facial acne scars

ELIGIBILITY:
Inclusion Criteria:

* Intent to undergo treatment of depressed acne scars
* Presence of 5-20 scars with a diameter of up to approximately 4 mm within the treatment area
* Similar type, size and number of scars on both cheeks
* Men or non-pregnant, non-breast feeding women
* Fitzpatrick skin type I-IV
* Signed and dated informed consent to participate in the study

Exclusion Criteria:

* Presence of more than 3 scars per cheek (within the treatment area) of the following types: icepick scars or atrophic acne scars with a diameter of > 4 mm.
* Active acne with inflammatory component
* Use of per oral or topical (facial) substances containing retinoids, bensoyl peroxide, alpha-hydroxy acid at concentrations above 10%, beta-hydroxy acid at a concentration above 2%, or antibiotic treatment for active acne within 4 months before treatment
* Use of isotretinoin within 6 months before treatment
* Post-surgical scars in the treatment area
* Previous tissue augmenting therapy or contouring with permanent filler or fat-injection in the treatment area
* Previous tissue augmenting therapy, contouring or revitalisation treatment with Calcium Hydroxyapatite (CaHa), or Poly L-Lactic Acid (PLLA), in the treatment area within 24 months before treatment
* Previous tissue augmenting therapy, contouring or revitalisation treatment with non-permanent filler such as hyaluronic acid (HA) or collagen in the treatment area within 12 months before treatment
* Previous tissue revitalisation treatment with neurotoxin, laser or light, mesotherapy, chemical peeling or dermabrasion in the treatment area within 6 months before treatment
* Previous surgery including aesthetic facial surgical therapy, liposuction, or tattoo in the treatment area
* Any medical condition that, in the opinion of the treating Investigator, would make the subject unsuitable for inclusion (e.g. a chronic, relapsing or hereditary disease that may interfere with the outcome of the study)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 49 (Actual)
Dates: Start 2017-04-20 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Galderma R&D
Locations (2):
- Germany (2):
  - Darmstadt, Darmstadt
  - Munich, Munich

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Dierickx C, Larsson MK, Blomster S. Effectiveness and Safety of Acne Scar Treatment With Nonanimal Stabilized Hyaluronic Acid Gel. Dermatol Surg. 2018 Nov;44 Suppl 1:S10-S18. doi: 10.1097/DSS.0000000000001689. PMID 30358630

RESULTS

PARTICIPANT FLOW:
Groups:
- Split-face: Treatment/No-treatment Control: All participants were randomized to receive treatment in either right or left cheek. The other cheek was a no-treatment control.
Period: Overall Study
Arm/Group | Split-face: Treatment/No-treatment Control
Started | 49
Completed 3 Month Visit | 47
Completed | 43
Not Completed | 6
Not completed — Lost to Follow-up | 4
Not completed — Subject request | 2

BASELINE CHARACTERISTICS:
Arm/Group | Split-face: Treatment/No-treatment Control
Number analyzed (Participants) | 49
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.3 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39
  Male | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 48
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Germany | 49

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Lower Scar Severity in the Treated Cheek Compared to the Untreated Cheek
Description: Overall scar severity assessed by blinded evaluator.
Time Frame: Month 3
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Split-face: Treatment/No-treatment Control
Number analyzed (Participants) | 47
percentage of participants | 81 [67 to 91]

2. Secondary Outcome: Percentage of Participants Improved on the Global Aesthetic Improvement Scale (GAIS)
Description: Assessed by blinded evaluator
Time Frame: Month 1, Month 3
Population: 48 participants at Month 1, 47 participants at Month 3, due to withdrawal. Split-face design: overall 48 participants, with one treated cheek and one cheek as no-treatment control.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Units Other Than Participants: cheeks
Arm/Group | No-treatment Control | Treatment
Number analyzed (Participants) | 48 | 48
Number analyzed (cheeks) | 48 | 48
percentage of participants
  Month 1 | 0 [0 to 0] | 96 [86 to 100]
  Month 3: number analyzed (Participants) | 47 | 47
  Month 3: number analyzed (cheeks) | 47 | 48
  Month 3 | 6 [1 to 18] | 83 [69 to 92]

ADVERSE EVENTS:
Time Frame: 1 year, 7 months
Arm/Group | Split-face: Treatment/No-treatment Control
All-Cause Mortality (participants affected / at risk) | 0/49
Serious Adverse Events (participants affected / at risk) | 1/49
Other Adverse Events (participants affected / at risk) | 9/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Split-face: Treatment/No-treatment Control (N=49)
Worsening of spinal disc herniation (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Split-face: Treatment/No-treatment Control (N=49)
Influenza (Infections and infestations) | 3 (3)
Nasopharyngitis (Infections and infestations) | 8 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-27): https://cdn.clinicaltrials.gov/large-docs/84/NCT03127384/Prot_SAP_000.pdf